CLINICAL TRIAL: NCT07219641
Title: Radicle Clarity RPN: A Randomized, Double-Blind, Placebo-Controlled Study Assessing the Impact of Health and Wellness Products on Cognitive Function and Related Health Outcomes.
Brief Title: Radicle Clarity RPN: A Study Assessing the Impact of Health and Wellness Products on Cognitive Function and Related Health Outcomes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX_P_2406_RPN
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Function

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on their age, assigned sex at birth and health outcome score during enrollment, then randomized to one of the study arms. Each participant will have an equal chance of being assigned to any study arm.
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Control (Placebo Comparator): Clarity Product Placebo Control
  Interventions: Dietary Supplement: Clarity Product Placebo Control
- Active Product 1 (Experimental): Clarity Active Product 1
  Interventions: Dietary Supplement: Clarity Active Product 1
- Active Product 2 (Experimental): Clarity Active Product 2
  Interventions: Dietary Supplement: Clarity Active Product 2

INTERVENTIONS:
Dietary Supplement: Clarity Product Placebo Control — Participants will use their Clarity Product Placebo Control as directed for a period of 6 weeks.
  Arms: Placebo Control
Dietary Supplement: Clarity Active Product 1 — Participants will use their Clarity Active Product 1 as directed for a period of 6 weeks.
  Arms: Active Product 1
Dietary Supplement: Clarity Active Product 2 — Participants will use their Clarity Active Product 2 as directed for a period of 6 weeks.
  Arms: Active Product 2

SUMMARY:
Radicle Clarity RPN: A Randomized, Double-Blind, Placebo-Controlled Study Assessing the Impact of Health and Wellness Products on Cognitive Function and Related Health Outcomes.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants will (1) have the opportunity for meaningful improvement (at least 30%) in their primary health outcome and (2) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants for 7 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world.

ELIGIBILITY:
- Inclusion

Participants must meet all the following criteria:

* Adults, at least 21 years of age at the time of electronic consent, inclusive of all ethnicities, races, and gender identities.

  * Assigned sex at birth will determine sex-specific recruitment and surveys (male vs female) employed, when needed.
* Resides in the United States.
* Has the opportunity for at least 30% improvement in their primary health outcome.
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study.

  * Exclusion

Individuals who report any of the following during screening will be excluded from participation:

* Report being pregnant, trying to become pregnant, or breastfeeding.
* Unable to provide a valid US shipping address and mobile phone number.
* Reports current enrollment in another clinical trial.
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day).
* Unable to read and understand English.
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients.

  * NYHA Class III or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure.
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients.

  * Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, seizure medications, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOIs, or thyroid products.
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s) that may limit the effects of the study products.
* Lack of reliable daily access to the internet.

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function | 7 weeks
  Change in cognitive function: Difference in rates of change over time in cognitive function score as assessed by PROMIS Cognitive Function 8A (scale 8-40; where lower scores correspond to worse cognitive function)

SECONDARY OUTCOMES:
Change in fatigue | 7 weeks
  Change in fatigue: Difference in rates of change over time in fatigue score as assessed by Patient Reported Outcome Measurement System (PROMIS) Fatigue 8A (scale 8-40; where higher scores correspond to more severe fatigue)
Change in sleep-related impairment | 7 weeks
  Change in sleep-related impairment: Difference between rates of change over time in sleep score as assessed by PROMIS Sleep-Related Impairment 8a (scale 8-40; where the higher scores correspond to worse sleep)
Change in cognitive abilities | 7 weeks
  Change in cognitive abilities: Difference between rates of change over time in Cognitive Abilities score as assessed by PROMIS Cognitive Function - Abilities 8a (scale 8-40; where the higher scores correspond to better cognitive abilities)

OTHER OUTCOMES:
Minimal clinically important difference (MCID) in cognitive function | 7 weeks
  Minimal clinically important difference (MCID) in cognitive function: Likelihood of experiencing minimal clinically important difference in cognitive function score as assessed by PROMIS Cognitive Function 8A (scale 8-40; where lower scores correspond to worse cognitive function)
Minimal clinically important difference (MCID) in fatigue | 7 weeks
  Minimal clinically important difference (MCID) in fatigue: Likelihood of experiencing minimal clinically important difference in fatigue score as assessed by PROMIS Fatigue 8A (scale 8-40; where higher scores correspond to more severe fatigue)
Minimal clinically important difference (MCID) in sleep | 7 weeks
  Minimal clinically important difference (MCID) in sleep: Likelihood of experiencing minimal clinically important difference in sleep score, as measured by PROMIS Sleep-Related Impairment 8a (scale 8-40; where the higher scores correspond to worse sleep)
Minimal clinically important difference (MCID) in cognitive abilities | 7 weeks
  Minimal clinically important difference (MCID) in cognitive abilities: Likelihood of experiencing minimal clinically important difference in cognitive abilities score as assessed by PROMIS Cognitive Function - Abilities 8a (scale 8-40; where the higher scores correspond to better cognitive abilities)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hewlings, Principal Investigator — Radicle Science
Locations (1):
- Radicle Science Inc., Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Related Info — https://www.radiclescience.com